CLINICAL TRIAL: NCT07149181
Title: A Multicenter, Prospective, Real-world Study Comparing the Efficacy and Safety of Chemotherapy Combined With or Without Immunotherapy as Postoperative Adjuvant Regimens in Patients With Resectable Gastric Cancer/Adenocarcinoma of the Esophagogastric Junction After Radical Surgery
Brief Title: Comparing the Efficacy and Safety of Chemotherapy Combined With or Without Immunotherapy as Postoperative Adjuvant Regimens in Patients With Resectable Gastric Cancer/Adenocarcinoma of the Esophagogastric Junction After Radical Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zheng Guoliang, Vice Offices Director, Liaoning Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoGC-03; KY20250315 (Other: Liaoning Cancer Hospital & Institute)
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Gastric / Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOX or XELOX with immunotherapy (Experimental)
  Interventions: Drug: SOX plus PD-1 inhibitor
- SOX or XELOX (Active Comparator)
  Interventions: Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: SOX plus PD-1 inhibitor — SOX or XELOX plus PD-1 inhibitor
  Arms: SOX or XELOX with immunotherapy
Drug: SOX Chemotherapy — SOX or XELOX
  Arms: SOX or XELOX

SUMMARY:
This study is to evaluate the efficacy and safety of chemotherapy combined with or without immunotherapy as postoperative adjuvant regimens in patients with resectable gastric cancer/adenocarcinoma of the esophagogastric junction after radical surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender not restricted;
2. Subjects diagnosed with gastric cancer (GC) or gastroesophageal junction cancer (GEJC) through imaging and other examinations, and with histopathological diagnosis of adenocarcinoma;
3. HER2 overexpression or amplification results are negative;
4. After radical surgery treatment, the investigator assesses that further adjuvant treatment is necessary, and the adjuvant treatment plan must be the one specified in this protocol.

Exclusion Criteria:

1. Gastric cancer that is known to be squamous cell carcinoma, undifferentiated carcinoma, or of other tissue types, or gastric cancer that is adenocarcinoma mixed with other tissue types;
2. Within 3 months before adjuvant therapy, there was a significant clinically significant bleeding symptom or a clear bleeding tendency;
3. Within 6 months before adjuvant therapy, had suffered from intestinal obstruction and/or had clinical signs or symptoms of digestive tract obstruction, including incomplete obstruction related to the original disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding;
4. Within 5 years before starting adjuvant therapy, was diagnosed with a malignant tumor (excluding malignant tumors with low metastasis and mortality risks, such as: skin basal cell carcinoma or cervical carcinoma in situ that has been adequately treated);
5. Within 30 days before starting adjuvant therapy, had participated in other clinical studies and used study drugs containing active ingredients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Compare the differences in the DFS rates between the two groups of subjects, DFS (Disease-Free Survival, which is the time from the start of postoperative adjuvant therapy until the first occurrence of recurrent disease. | The observation period starts from the time the postoperative adjuvant therapy begins and lasts for at least 2 years

SECONDARY OUTCOMES:
Compare the differences in the OS rates between the two groups of subjects, OS (Overall Survival, which refers to the time from the start of postoperative adjuvant therapy until death due to any cause) | The observation period starts from the time the postoperative adjuvant therapy begins and lasts for at least 2 years
The Adverse Events of anti-PD1/PDL1 monoclonal antibody combined with chemotherapy versus chemotherapy in postoperative adjuvant treatment for gastric cancer/adenocarcinoma of the esophagogastric junction | The observation period starts from the time the postoperative adjuvant therapy begins and lasts for at least 2 years